CLINICAL TRIAL: NCT07228520
Title: Strength and Pain-Coping Through Resilience and Knowledge
Acronym: SPARK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00529967
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Pain; Depressive Symptoms; Aging
Keywords: Older Adults
MeSH Terms: conditions — Pain; Depression

STUDY DESIGN:
Intervention Model Description: The investigator will conduct subsequent single blind wait list control design to test the preliminary effects of DAPPER and the feasibility of older African American women integrating strategies to address pain, depression, and frailty that are tailored to the individual into the individual's daily routines.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The statistician will be responsible for randomization and the investigator and study team will not have knowledge if participants are assigned to intervention group or wait list control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPARK Intervention Arm (Experimental): The intervention group will receive the intervention for 12 weeks. The wait list control group will have outcomes measured but will not receive the intervention at this time.
  Interventions: Behavioral: SPARK
- Wait List Control Arm (Active Comparator): Once the intervention group has completed the intervention the wait list control group will complete the intervention.
  Interventions: Behavioral: SPARK

INTERVENTIONS:
Behavioral: SPARK — The SPARK program is person directed and will consist of 8 nurse visits during which the nurse assesses each participant for pain, depression and frailty and then implements a manualized individually tailored intervention. Participants will be randomized into either the intervention or the wait list control group. Once the intervention group has completed the intervention group's visits, the wait list control group will begin the waitlist control group's visits. All participants will all be offered the same information and format of nurse visits. The nurses will systematically tailor the content of the visits to the participants' risk profile and goals based on protocols. All participants will be assessed at the start of the study, at 12 weeks and 24 weeks.

SUMMARY:
Older adults who are 50 years of age and older with depressive symptoms, pain and difficulty with mobility will participate in the SPARK intervention study that includes 8 nurse visits in participants' homes to help participants with participants' pain and mood.

DETAILED DESCRIPTION:
SPARK (Strength and Pain-Coping through Resilience and Knowledge) is a home-based, nurse-delivered behavioral intervention designed to reduce pain interference and depressive symptoms among community-dwelling older adults with mobility limitations. Chronic pain and depression occurs together later in life and can impair daily function, independence, and overall well-being. Pain interference, how pain affects daily life, is a critical and actionable outcome that is closely linked to depressive symptoms. SPARK integrates evidence-informed strategies delivered through the Neighborhood Nursing model and brings the necessary care directly to the homes of the participants. The intervention comprises eight weekly individualized 1:1 nurse home visits that integrate goal-directed care planning, education on pain and mood self-management, and coordination with Neighborhood Nursing and Community Health workers to address barriers and leverage local resources.

ELIGIBILITY:
Inclusion Criteria:

* Self-report pain >3 out of a 0 -10 scale that has lasted longer than 3 months and keeps subjects from doing at least one activity that subjects would like to do
* Live in the community
* Live in Central Maryland
* Score a 5 or higher on the PHQ-9 (depression measure) at least two times during a two week period (screening call and then at first data collection visit)
* Must be pre-frail (one or two criteria on frailty phenotype) or frail (three or more of the criteria on frailty phenotype)
* One ADL or IADL limitation

Exclusion Criteria:

* Hospitalized > 3 times in the last year
* Participating in physical therapy
* Have a terminal diagnosis (<1 year expected survival)
* > moderate intellectual impairment (5-7 errors) based on the Short Portable Mental Status Questionnaire (SPMSQ)
* Unable to speak or understand English

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity as assessed by the Patient Reported Outcomes Measurement Information System (PROMIS) | Baseline, 12 weeks and 24 weeks
  The PROMIS Intensity is used to measure pain intensity on a scale of 0-10. Higher scores indicate more pain intensity.
Change in Pain Interference as assessed by the PROMIS Pain Interference | Baseline, 12 weeks and 24 weeks
  The Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference is a six item scale used to measure how much pain interferes with activities. The scores can range from 6-30. Higher scores indicate more pain interference with activities.
Change in Depressive Symptoms as assessed by the Patient Health Questionnaire 9 (PHQ-9) | Baseline, 12 weeks and 24 weeks
  The Patient Health Questionnaire 9 (PHQ-9) includes 9 questions related to the Diagnostic and Statistical Manual of Mental Disorders (DSM) diagnostic criteria for major depression. The PHQ-9 scores range from 0-27. Higher scores indicate more depressive symptoms.
Change in Depressive Symptoms as assessed by the PROMIS 57 | Baseline, 12 weeks and 24 weeks
  The Patient Reported Outcomes Measurement System (PROMIS)57 the Patient Reported Outcomes Measurement Information System (PROMIS) 57, which is includes an 8-item instrument that can be used to measure self-reported negative mood, view of self, and somatic symptoms. The score range for PROMIS 57 is 8-40. Higher scores indicate more depressive symptoms.

SECONDARY OUTCOMES:
Change in Physical Function as assessed by the Katz Activities of daily living (ADL) | Baseline, 12 weeks and 24 weeks
  The Katz Activities of daily living (ADL) is used measure physical function through ability to perform activities of daily living. Score ranges are from 0-6 with 6 indicating full function and a score of 2 or less indicating severe functional impairment.
Change in Physical Function as assessed by the Lawton's Instrumental Activities of Daily Living (IADL) | Baseline, 12 weeks and 24 weeks
  Lawton's Instrumental Activities of Daily Living (IADL) measures instrumental activities of daily living as a measure of physical function. The scores range from 0-8 with higher scores indicating better physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Janiece L Taylor, PhD, Principal Investigator — Johns Hopkins School of Nursing; Catherine Clair, MHS, Study Director — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor JL, Clair CA, Lee JW, Atkins S, Riser TJ, Szanton SL, McCoy MC, Thorpe RJ Jr, Wang C, Gitlin LN. A protocol for a wait list control trial of an intervention to improve pain and depressive symptoms among middle-aged and older African American women. Contemp Clin Trials. 2023 Sep;132:107299. doi: 10.1016/j.cct.2023.107299. Epub 2023 Jul 20. PMID 37478967
- [Result] Taylor JL, Clair CA, Gitlin LN, Atkins S, Bandeen-Roche K, Abshire Saylor M, Hladek MD, Riser TJ, Thorpe RJ Jr, Szanton SL. Acceptability and Feasibility of a Pain and Depressive Symptoms Management Intervention in Middle-Aged and Older African American Women. Innov Aging. 2023 Sep 8;7(10):igad096. doi: 10.1093/geroni/igad096. eCollection 2023. PMID 38094930
- Available data/document: Study Protocol: 37478967 — https://pubmed.ncbi.nlm.nih.gov/37478967/
- Available data/document: Outcomes Manuscript: 38094930 — https://pubmed.ncbi.nlm.nih.gov/38094930/